CLINICAL TRIAL: NCT07084870
Title: HIGH FLOW NASAL OXYGEN VERSUS BILEVEL POSITIVE AIRWAY PRESSURE VENTILATION IN PREECLAMPTIC PATIENTS WITH ACUTE HYPOXAEMIC RESPIRATORY FAILURE
Brief Title: HFNO VERSUS BIPAP IN PREECLAMPTIC PATIENTS WITH ACUTE HYPOXAEMIC RESPIRATORY FAILURE
Acronym: HFNO BIPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0201403
Record Dates: First submitted 2025-07-23; First posted 2025-07-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HFNO vs BIPAP; Preeclamptic Acute Hypoxaemic Respiratory Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): 30 preeclamptic patients with acute hypoxaemic respiratory failure who received O2 therapy via HFNC
  Interventions: Other: High flow nasal oxygen
- Group 2 (Experimental): 30 preeclamptic patients with acute hypoxaemic respiratory failure who received non-invasive BiPAP ventilation.
  Interventions: Other: non invasive BIPAP

INTERVENTIONS:
Other: High flow nasal oxygen — Patients in group I then received HFNO. The initial flow rate was adjusted to 50L/min and gradually reduced as tolerated by the patient. The humidification chamber temperature was set at 37°C and gradually reduced to the patient comfort. FiO2 was 100% and then gradually reduced over time according to improvement in oxygenation.
  Arms: Group 1
Other: non invasive BIPAP — Patients in group II received oxygen therapy via intermittent non- invasive positive pressure ventilation, BiPAP mode ventilator using a face mask. BiPAP settings were adjusted as follows: P (low) of 5cm H2O to 10cm H2O and an inspiratory pressure P (high) of 10-20cm H2O . FiO2 was adjusted to 100% and then gradually reduced over time according to improvement in oxygen saturation and PaO2/Fio2 ratio. Respiratory rate was adjusted from 10-12 at then changed according to patient´s respiratory effort and according to ABG.
  Arms: Group 2

SUMMARY:
The aim of this study was to evaluate the use of HFNO to support oxygenation in acute hypoxemic respiratory failure in postpartum pre-eclamptic patients, compared with non-invasive intermittent bilevel positive airway pressure ventilation

DETAILED DESCRIPTION:
Patients in group I will receive HFNO by AIRVO™ (Fisher & Paykel Healthcare Ltd., Auckland, New Zealand). The initial flow rate will be 50L/min and will eventually be diminished in case of intolerance. Humidification chamber temperature will be set at 37 °C and will eventually be diminished in case of intolerance. FiO2 will be 100% and then gradually reduced to 50% when pulse oximetry values are acceptable. Patients in the group II will receive oxygen therapy via intermittent non- invasive positive pressure ventilation, BiPAP mode Dräger Savina ventilator, and a face mask will be used. P (low) of 5 cm H2O to 10 cm H2O and an inspiratory pressure P (high) of 10-20 cm H2O above PEEP. FiO2 will be 100% and then gradually reduced to 50 % when pulse oximetry values are acceptable. Respiratory rate will be from 10-12. It will be applied for 30 minutes every hour with 30 minutes rest, and will be applied continuously for 6-8 hours at night. The size of the face mask will be chosen to optimize subject comfort while minimizing air leaks. If the patient cannot tolerate the treatment, she will be excluded from the study. Patients will be assessed for treatment weaning then interruption when they meet the following criteria:

* Respiratory rate ≤24 breaths/min
* No recruitment of accessory muscles of respiration during calm breathing.
* Haemodynamic stability (heart rate <110/min; mean blood pressure between 60 and 90 mmHg and no Haemodynamically significant arrhythmias.
* SpO2 > 95 % on FIO2 ≤30.
* Improvement of blood gases.

Criteria for treatment failure and the need for intubation:

* Respiratory rate > 25 breaths/min
* The use of accessory muscles of respiration.
* Haemodynamic instability (heart rate >110/min; mean blood pressure below 90 or significant arrhythmias.
* Failure to achieve SpO2 above 91.
* PaO2/ FiO2 ratio <150, PaCO2 >45 or PH <7.30.

ELIGIBILITY:
Inclusion Criteria:

preeclamptic postpartum patients, admitted to obstetric intensive care unit (ICU) due to acute hypoxaemic respiratory failure, fully conscious with The American Society of Anesthesiologists (ASA) class II or III.

Exclusion Criteria:

1. Patients with PaCO2 more than 45 mmHg.
2. Unconscious patients.
3. PaO2/ FiO2 ratio less than 150.
4. Known cardiac disease.
5. Hemodynamic instability.
6. Facial deformity.
7. Morbid obese patients with BMI >40

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postpartum preeclamptic patients
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
treatment success | 48 hours
  measure the success of treatment technique by the improvement of PaO2/ FiO2 ratio, peripheral oxygen saturation
Treatment failure | 48 hours
  reatment failure by recording the number of tracheal intubations in the first 48 hours after the start of the treatment

SECONDARY OUTCOMES:
Assess the level of oxidative stress by measuring serum level of soluble Nox2 derived peptide (sNOX2-dp), a marker of NADPH-oxidase activation | 6 hours
  Extracellular levels of soluble NOX2 derived peptide (sNOX2-dp), a marker of NADPH oxidase activation, will be detected by ELISA. It will be measured on admission and 6 hours after initiation of oxygen therapy
Assess the patient's comfort and tolerance to the technique used. | 48 hours
  assessed by Visual numeric scale (VNS): A range from 1 to 5 will be used. With 1 very comfortable,2 comfortable, 3 uncomfortable, 4 very uncomfortable, 5 the worst discomfort.
Record any possible complications related to treatment. Record any possible complications related to treatment. Record any possible complications | 48 hours
  Record any possible complications related to treatment.
  Facial skin erythema, nasal skin lesions, eye irritation, vomiting related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shahira Ahmed Yousef Elmetiny, MD, Study Director — Alexandria University; Tarek Atef Tawfik, MD, Study Director — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
through clinical trials
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: HFNO, BIPAP, acute hypoxaemic respiratory failure, preeclampsia